CLINICAL TRIAL: NCT01636765
Title: Study of Inter- and Intra-rater Reliability of the Clinician Erythema Assessment Scale
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 199201-003
Record Dates: First submitted 2012-07-09; First posted 2012-07-10 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Erythema; Rosacea
MeSH Terms: conditions — Erythema; Rosacea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Patients with facial erythema associated with rosacea. There was no intervention in this study.
  Interventions: Drug: No Intervention

INTERVENTIONS:
Drug: No Intervention — No intervention.

SUMMARY:
This is a study to evaluate inter- and intra-rater reliability of the Clinician Erythema Assessment Scale. There is no treatment (intervention) associated with this study.

ELIGIBILITY:
Inclusion Criteria:

* Rosacea

Exclusion Criteria:

* Unwilling to remove all facial make-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with facial erythema related to rosacea
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 104
Completed | 104
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 104
Age, Continuous [Mean (Full Range); unit: Years] | 44.2 [19 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Inter-rater Reliability of the Clinician Erythema Assessment (CEA) Scale
Description: Inter-rater agreement (among raters) of the CEA scores (0=clear skin with no signs of erythema; 1=almost clear of erythema, slight redness; 2=mild erythema, definite redness; 3=moderate erythema, marked redness; 4=severe erythema, fiery redness) evaluated using Kendall's coefficient of concordance (Kendall's W). Each of 7 raters scored 104 participant's severity of erythema due to rosacea using the CEA Scale at 2 different time points at day 1. The overall inter-rater agreement for Kendall's W for all raters combined was estimated based on the average of the scores from those 2 different time points. The degree of agreement of the point estimates of Kendall's W was interpreted according to the reference range scale that was pre-defined as: ≤ 0=poor, 0.00-0.20=slight, 0.21-0.40=fair, 0.41-0.60=moderate, 0.61-0.80=substantial and 0.81-1.00=almost perfect. The 95% confidence interval for Kendall's W was provided.
Time Frame: Day 1
Population: All enrolled participants.
Measure: Mean (95% Confidence Interval); unit: Kendall's W
Arm/Group | All Participants
Number analyzed (Participants) | 104
Kendall's W | 0.908 [0.703 to 1.000]

2. Primary Outcome: Intra-rater Reliability of the CEA Scale
Description: Intra-rater (within raters) agreement of the CEA scores (0=clear skin with no signs of erythema; 1=almost clear of erythema, slight redness; 2=mild erythema, definite redness; 3=moderate erythema, marked redness; 4=severe erythema, fiery redness) was evaluated by weighted Kappa statistics (WKS). WKS were calculated for each of 7 raters who evaluated 104 participant's severity of erythema of rosacea using the CEA scale, assessing agreement between 2 different time points at day 1. The overall intra-rater agreement for WKS for all raters combined was estimated by pooling WKS for each rater using a chi-square statistic. The degree of agreement of the point estimates of WKS was interpreted according to the reference range scale that was predefined as: ≤ 0=poor, 0.00-0.20=slight, 0.21-0.40=fair, 0.41-0.60=moderate, 0.61-0.80=substantial and 0.81-1.00=almost perfect. The 95% confidence interval for Kappa statistics was provided.
Time Frame: Day 1
Population: All enrolled participants.
Measure: Mean (95% Confidence Interval); unit: Kappa statistics
Arm/Group | All Participants
Number analyzed (Participants) | 104
Kappa statistics | 0.752 [0.722 to 0.783]

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/104
Other Adverse Events (participants affected / at risk) | 0/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.